CLINICAL TRIAL: NCT00360997
Title: Mobilisation and Tactile Stimulation to Enhance Upper Limb Recovery After Stroke: Phase I Investigation of Acceptable Dose, Efficacy and Underlying Mechanisms
Brief Title: Investigation of Acceptable Dose of Mobilisation and Tactile Stimulation to Enhance Upper Limb Recovery After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSA 2005/03
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Stroke
Keywords: Stroke rehabilitation; Physical therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioural (Other): Conventional UK physical therapy (Con UK PT)
  Interventions: Behavioral: Conventional UK physical therapy
- Con UK PT + MTS (Experimental): Con UK PT + 30/60 or 120 minutes MTS
  Interventions: Procedure: Con UK PT + Mobilisation & tactile stimulation (MTS)

INTERVENTIONS:
Behavioral: Conventional UK physical therapy
  Other Names: Con UK PT
  Arms: Behavioural
Procedure: Con UK PT + Mobilisation & tactile stimulation (MTS) — Con UK PT + Mobilisation & Tactile Stimulation (MTS) which is further randomised to 30, 60 or 120 mins/day
  Other Names: Con UK PT + MTS
  Arms: Con UK PT + MTS

SUMMARY:
The purpose of this study is to find which of three doses of mobilisation and tactile stimulation therapy, when given in addition to conventional UK physical therapy, has the most beneficial effect on enhancing motor recovery of the upper limb early after stroke.

DETAILED DESCRIPTION:
Background The scientific evidence indicates that upper limb motor recovery may be enhanced with the appropriate dose of afferent stimulation normally arising from functional activities. Even if the appropriate dose was known, people with severe paresis or paralysis would not be able to participate in functional training. For these people "mobilization and tactile stimulation" (MTS) therapy might enhance: upper limb recovery, and, changes in brain regions that can influence motor output.

Questions In stroke patients with paralysis or severe paresis which dose of MTS therapy a) produces the least adverse events; b) has the most beneficial effect on voluntary muscle contraction and functional ability. This study will also address: c) whether the magnitude of sensory/motor cortex activation prior to MTS can predict response to MTS; and, d) whether changes in sensory and/or motor cortex activation correlate with improvement.

Subjects (n=80) from two clinical centres with an anterior cerebral circulation stroke 8 to 84 days before recruitment, paresis or severe paralysis and no clinically important pain affecting the upper arm or shoulder after stroke.

Methods After baseline measures (Day 1) subjects will be randomised to a) no extra therapy; or one of three doses of MTS therapy for 14 consecutive working days, b) 30 minutes; c) 60 minutes; or, d) 120 minutes. All subjects will receive the conventional therapy normally provided within each centre. On Day 16, outcome measures will be made. The experimental intervention, MTS therapy will be individualised for each subject from a standardised schedule of techniques within treatment categories including: passive movements, massage; specific sensory input; and, functional movement. The measurement battery will be: a) efficacy, Motricity Index Arm Section and the Action Research Arm Test; b) adverse events, presence of upper limb pain and decrease in Motricity Index score; and c) Functional MRI (London subjects), T1 weighted anatomical images and T2* weighted MRI transverse echo-planar images undertaking these studies with both sensory and motor paradigms where feasible.

Analysis Analysis for efficacy and adverse events will be conducted using the Chi-squared test for trend or linear regression as appropriate. The results will be combined to determine the most appropriate dose of MTS. Imaging data will be processed using Statistical Parametric Mapping and then analysed statistically using a least mean squares fit of the model to the data to determine regions of significant activation for each session.

ELIGIBILITY:
Inclusion Criteria:

* Have suffered an infarct or haemorrhage in the anterior cerebral circulation, confirmed by neuroimaging, 8 to 84 days before recruitment
* Have a paralysed or severely paretic upper limb as measured by a score of 61/100 or less on the Motricity Index Arm Section17

Exclusion Criteria:

* Clinically important pain affecting the upper arm or shoulder when recruited to this study
* Visible upper limb movement deficits attributable to pathology other than stroke
* Unable to follow a 1-stage command using their non-paretic upper limb (ie severe communication or other cognitive deficits precluding ability to participate in MTS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Efficacy: Primary outcome, Motricity Index - arm

SECONDARY OUTCOMES:
Efficacy: Action Research Arm Test (ARAT).
Adverse events: Occurrence of upper limb pain and decrease Motricity score
Underlying mechanisms: Functional MRI for suitable London subjects
Underlying mechanisms: Transcranial magnetic stimulation to measure evoked motor potentials in paretic upper limb for suitable London subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Valerie M Pomeroy, PhD, Study Chair — St George's, University of London
Locations (2):
- United Kingdom (2):
  - North Staffordshire Combined Healthcare NHS Trust, Stoke-on-Trent, Staffordshire
  - St Thomas' Foundation Hospital NHS Trust, London